CLINICAL TRIAL: NCT03265145
Title: Randomized Pragmatic Clinical Trial in a Community-Based Setting Comparing STIOLTO® RESPIMAT® vs. ICS-LABA Plus LAMA in Patients With COPD
Brief Title: Assessment In a Real World Setting of the Effect of Inhaled Steroid-based Triple Therapy Versus the Combination of Tiotropium and Olodaterol on Reducing Chronic Obstructive Pulmonary Disease (COPD) Exacerbations [AIRWISE]
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Carelon Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1237-0064
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; laminin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stiolto Respimat (Experimental)
  Interventions: Drug: Stiolto Respimat
- ICS plus LABA plus LAMA (triple therapy) (Active Comparator): ICS (Inhaled Corticosteroid) plus LABA (Long-Acting Beta Agonist) plus (Long-Acting Muscarinic Antagonist)
  Interventions: Drug: ICS (Inhaled Corticosteroid) (Triple therapy); Drug: LABA (Long-Acting Beta Agonist) (Triple therapy); Drug: LAMA (Long-Acting Muscarinic Antagonist) (Triple therapy)

INTERVENTIONS:
Drug: Stiolto Respimat — Duration - 12 months
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO
  Arms: Stiolto Respimat
Drug: ICS (Inhaled Corticosteroid) (Triple therapy) — Duration - 12 months
  Arms: ICS plus LABA plus LAMA (triple therapy)
Drug: LABA (Long-Acting Beta Agonist) (Triple therapy) — Duration - 12 months
  Arms: ICS plus LABA plus LAMA (triple therapy)
Drug: LAMA (Long-Acting Muscarinic Antagonist) (Triple therapy) — Duration - 12 months
  Arms: ICS plus LABA plus LAMA (triple therapy)

SUMMARY:
The primary objective of this pragmatic study is to compare the time to first moderate or severe COPD exacerbation in patients, not controlled on their current therapy, randomized to Stiolto Respimat versus triple therapy over 12 months of treatment

The secondary objectives of this study include:

1. To compare the annual rate of moderate or severe COPD exacerbations for patients on Stiolto Respimat with patients on triple therapy.
2. To compare the time to first severe COPD exacerbation in both treatment arms.
3. To compare the annual rate of severe COPD exacerbations in both treatment arms.
4. To compare the proportion of patients with moderate or severe COPD exacerbations in both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis as defined by the study physician
* Currently on one of the following maintenance therapies:

  * LAMA monotherapy
  * LABA monotherapy
  * ICS/LABA (FDC)
* Physician determination that patient is not controlled on current pharmacotherapy
* Adult patient 40 years of age or older at time of study enrollment
* Willingness and ability to understand and provide documented Informed Consent Form (ICF) and Health Insurance Portability and Accountability Act (HIPAA) Authorization Form prior to commencement of any study required assessments, either directly or through Legally Authorized Representative.

Exclusion Criteria:

* Currently on LAMA/LABA (free or FDC) or triple therapy (ICS plus LABA plus LAMA)
* Contraindication to any study medications (LAMA, LABA or ICS)
* Documented diagnosis of current asthma
* Pregnant or nursing women
* Women of childbearing potential are not restricted in this trial, however it is expected that the investigator will assess the risks and benefits of the assigned treatment as per the product label(s) and discuss this with any women of childbearing potential prior to providing the patient with the prescription for the assigned treatment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (89):
- United States (89):
  - Pulmonary Associates of Mobile, PC, Mobile, Alabama
  - Healthscan Clinical Trials LLC, Montgomery, Alabama
  - HealthScan Research, Montgomery, Alabama
  - Diamond Childrens Medical Center, Tucson, Arizona
  - CareMore Apple Valley Care Center, Apple Valley, California
  - HealthCare Partners, Commerce, California
  - Advanced Research Center, Inc., Murrieta, California
  - Newport Native MD, Inc, Newport Beach, California
  - Aureus Medical Group, Inc, Rancho Cucamonga, California
  - Capital Allergy and Respiratory Disease Center, Roseville, California
  - Paloma Medical Group, San Juan Capistrano, California
  - Adnab Research/Prestige Care Physician, Torrance, California
  - Pulmonary and Sleep of Tampa Bay, Brandon, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Saint Francis Sleep, Allergy and Lung Institute, LLC, Clearwater, Florida
  - Cohen Medical Research Associates, LLC, Delray Beach, Florida
  - Gary J. Richmond, M.D., PA, Fort Lauderdale, Florida
  - Medical Research of Central Florida, Leesburg, Florida
  - Florida Lung and Sleep Associates, Lehigh Acres, Florida
  - TRY Research, Maitland, Florida
  - Pro Live Medical Research, Miami, Florida
  - Advanced Research for Health Improvement, LLC, Naples, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - Bassetti Medical Research Inc, Sebring, Florida
  - Pasadena Ctr for Medical Rsrch, St. Petersburg, Florida
  - John Suen MD PA, Vero Beach, Florida
  - Gwinnett Research Institute, Buford, Georgia
  - Pulmonary and Sleep Specialists, PC, Decatur, Georgia
  - DC Pulmonary Medicine, Marietta, Georgia
  - Southern IL Clinical Rsrch Ctr, O'Fallon, Illinois
  - American Health Network of Indiana, LLC, Franklin, Indiana
  - American Health Network of Indiana, LLC, Greenfield, Indiana
  - The LaPorte County Institute for Clinical Research, Michigan City, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - American Health Network, New Albany, Indiana
  - Kentucky Lung Clinic, Georgetown, Kentucky
  - Pulmonary and Sleep Clinic PLLV, Hopkinsville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Pulmonary and Critical Care Associates of Baltimore, Bel Air, Maryland
  - Pulmonary and Critical Care Associates of Baltimore, Towson, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Vida Clinical Studies, Dearborn, Michigan
  - Flint Clinical Research, Flint, Michigan
  - Mercy Surgery Center, Springfield, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - Jubilee Clinical Research, Inc, Las Vegas, Nevada
  - Shore Pulmonary, PA, Ocean City, New Jersey
  - Bassett Medical Center, Cooperstown, New York
  - Pulmonary Health Physicians, Fayetteville, New York
  - Feinstein Institute for Medical Research, New Hyde Park, New York
  - Lenox Hill Hospital, New York, New York
  - Orchard Park Family Practice, Orchard Park, New York
  - American Health Research, Inc., Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Coastal Carolina Health Care, P.A., New Bern, North Carolina
  - Tabor City Family Medicine, Tabor City, North Carolina
  - Goshen Medical Center, Whiteville, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Catherine LaRuffa, MD, Inc., Blanchester, Ohio
  - Valley Medical Primary Care, Centerville, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Midwest Pulmonary and Sleep Research, Dayton, Ohio
  - Ohio Sleep and Pulmonary Center, Englewood, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Robert Santiago MD, Inc., Galion, Ohio
  - Pulmonary, Critical Care and Sleep Medicine Associates, Hamilton, Ohio
  - Wells Inst for Hlth Awareness, Kettering, Ohio
  - Pulmonary Medicine, South Euclid, Ohio
  - Toledo Clinic Incorporated, Toledo, Ohio
  - Ohio Clinical Research, LLC, Willoughby Hills, Ohio
  - Comprehensive Internal Medicine, Inc., Wooster, Ohio
  - Preferred Primary Care Phys, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Frontier Clinical Research LLC, Smithfield, Pennsylvania
  - Preferred Primary Care Phys, Uniontown, Pennsylvania
  - Carolina Medical Research, Clinton, South Carolina
  - Main Street Physicians Care, Little River, South Carolina
  - Family Medicine of SayeBrook, Myrtle Beach, South Carolina
  - Houston Pulmonary Sleep Allergy and Asthma Associates, Cypress, Texas
  - Texas Health Physicians Group, Dallas, Texas
  - North Texas Lung & Sleep Clnc, Fort Worth, Texas
  - SMS Clinical Research, Mesquite, Texas
  - San Marcos Family Medicine, San Marcos, Texas
  - Texarkana Clinical Research, Texarkana, Texas
  - Chesapeake Pulmonary and Critical Care, Chesapeake, Virginia
  - Richmond Family Practice, Richmond, Virginia
  - MultiCare Institute, Cheney, Washington
  - Western Washington Medical Grp, Everett, Washington
  - Pulmonary and Critical Care Associates, SC, Cudahy, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a pragmatic randomized open label active controlled parallel group design trial conducted in a real-world, community-based practice setting. Participants were on long-acting muscarinic antagonist (LAMA), long-acting beta agonist (LABA) or Inhaled Corticosteroid (ICS)/LABA for COPD, but were determined by their physician to not be controlled on their current therapy. Subjects were randomized to either Stiolto Respimat or ICS plus LABA plus LAMA (triple therapy) for the study.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Stiolto® Respimat®: Patients with chronic obstructive pulmonary disease (COPD) who were on long-acting muscarinic antagonist (LAMA) or long-acting beta agonist (LABA) or inhaled corticosteroid (ICS)/LABA maintenance therapy, and whose treatment was not controlled on the medication regimen as determined by the physician.
  Patients started the following Stiolto® Respimat® treatment: Fixed dose of 2.5 micrograms (mcg) tiotropium and 2.5 mcg olodaterol (Stiolto® Respimat®) per actuation were inhaled twice daily (tiotropium/olodaterol daily dosage: 5/5 mcg). Patients were followed for 12 months regardless of treatment switching or discontinuing study treatment.
- ICS Plus LABA Plus LAMA (Triple Therapy): Patients with chronic obstructive pulmonary disease (COPD) who were on long-acting muscarinic antagonist (LAMA) or long-acting beta agonist (LABA) or inhaled corticosteroid (ICS)/LABA maintenance therapy, and whose treatment was not controlled on the medication regimen as determined by the physician.
  Patients started the following ICS plus LABA plus LAMA (triple therapy) treatment made up of the combination of any approved drugs that their physician chooses.Triple Therapy (ICS + LABA + LAMA) was inhaled with dose as prescribed by physicians per label for selected medications. Patients were followed for 12 months regardless of treatment switching or discontinuing study treatment.
Period: Overall Study
Arm/Group | Stiolto® Respimat® | ICS Plus LABA Plus LAMA (Triple Therapy)
Started | 356 | 358
Completed (12 Month Study Observation Period) | 285 | 302
Not Completed | 71 | 56
Not completed — Protocol Violation | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 23 | 19
Not completed — Death | 12 | 12
Not completed — Lost to Follow-up | 13 | 9
Not completed — missing end of study form, could not definitely count as completion or discontinuation | 0 | 1
Not completed — Switched back to previous medication | 1 | 0
Not completed — Did not want to take medication | 1 | 0
Not completed — Subject could not afford medication | 0 | 1
Not completed — Site closed | 2 | 3
Not completed — Incorrectly randomized | 16 | 6
Not completed — Entered into Electronic Data Capture in error | 0 | 1
Not completed — Physician Decision | 0 | 3
Not completed — Subject transferred to another facility | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population: The ITT population will include all randomized patients allocated to their original randomized treatment group, even if they switched or discontinued study treatment. Due to investigator error, 5 patients in each group received the prescription for the wrong treatment. These subjects were included in the actual treatment, not the randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stiolto® Respimat® | ICS Plus LABA Plus LAMA (Triple Therapy) | Total
Number analyzed (Participants) | 356 | 358 | 714
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (9.32) | 69.9 (9.81) | 69.5 (9.57)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 181 | 174 | 355
  Female | 169 | 181 | 350
  Missing | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 20 | 40
  Not Hispanic or Latino | 329 | 334 | 663
  Unknown or Not Reported | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 292 | 300 | 592
  Black or African American | 42 | 38 | 80
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 9 | 9 | 18
  Missing | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time to First Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Over the 12 Month Study Period
Description: Time to first moderate or severe chronic obstructive (COPD) exacerbation over 12 months of treatment pulmonary disease.
  Moderate exacerbation was a patient receiving an exacerbation-related prescription such as oral corticosteroid (prednisone or prednisolone) and/or antibiotic, but not requiring hospitalization.
  Severe exacerbation was a patient requiring hospitalization or emergency room visit due to COPD (ICD-9-491.21 or ICD-10-J44.1).
  Median survival time as well as 95% confidence interval was calculated using Kaplan-Meier curves.
Time Frame: Baseline till end of study, up to 12 months.
Population: Intent to Treat (ITT) Population: The ITT population will include all randomized patients allocated to their original randomized treatment group, even if they switched or discontinued study treatment. Only patients with non missing ICS baseline values were included. Due to investigator error, 5 patients in each group received the prescription for the wrong treatment. These subjects were included in the actual treatment, not the randomized treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stiolto® Respimat® | ICS Plus LABA Plus LAMA (Triple Therapy)
Number analyzed (Participants) | 348 | 354
Months | NA [NA to NA] — Non-calculable as the median was not reached (and neither was the Q1). | NA [NA to NA] — Non-calculable as the median was not reached (and neither was the Q1).
Statistical Analysis 1: Comparison: Stiolto® Respimat® vs ICS Plus LABA Plus LAMA (Triple Therapy); Test type: Other; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.87 to 1.72] — Cox proportional hazards model with baseline ICS prior use as a covariate was used to estimate the hazard ratio (HR) and the two-sided 95% Wald confidence interval (CI). Ratio: Stiolto Respimat/triple therapy

2. Secondary Outcome: Annual Rate of Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: Annual rate of moderate or severe chronic obstructive pulmonary disease (COPD) exacerbations.
  Moderate exacerbation was a patient receiving an exacerbation-related prescription such as oral corticosteroid (prednisone or prednisolone) and/or antibiotic, but not requiring hospitalization.
  Severe exacerbation was a patient requiring hospitalization or emergency room visit due to COPD (ICD-9-491.21 or ICD-10-J44.1).
  Annual rate analysis utilized a negative binomial model with fixed effect of treatment (Stiolto Respimat versus triple therapy), logarithm of observational time as offset, and baseline prior ICS was used as a covariate.
Time Frame: Baseline till end of study, up to 12 months.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Groups:
- Triple Therapy: Patients with chronic obstructive pulmonary disease (COPD) who were on long-acting muscarinic antagonist (LAMA) or long-acting beta agonist (LABA) or inhaled corticosteroid (ICS)/LABA maintenance therapy, and whose treatment was not controlled on the medication regimen as determined by the physician.
  Patients were switched to a treatment of ICS plus LABA plus LAMA (triple therapy), made up of the combination of any approved drugs that their physician chooses, for 12 months of treatment.
Arm/Group | Stiolto® Respimat® | Triple Therapy
Number analyzed (Participants) | 348 | 354
Exacerbations per participant per year | 0.36 [0.28 to 0.47] | 0.26 [0.19 to 0.34]
Statistical Analysis 1: Comparison: Stiolto® Respimat® vs Triple Therapy; Test type: Other; adjusted annual rate ratio = 1.41, 95% CI 2-sided [0.97 to 2.04] — Ratio: Stiolto Respimat/triple therapy

3. Secondary Outcome: Time to First Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Over 12 Months of Treatment Pulmonary Disease
Description: Time to first severe chronic obstructive (COPD) exacerbation over 12 months of treatment pulmonary disease.
  Moderate exacerbation was a patient receiving an exacerbation-related prescription such as oral corticosteroid (prednisone or prednisolone) and/or antibiotic, but not requiring hospitalization.
  Severe exacerbation was a patient requiring hospitalization or emergency room visit due to COPD (ICD-9-491.21 or ICD-10-J44.1).
  Median survival time as well as 95% confidence interval was calculated using Kaplan-Meier curves.
Time Frame: Baseline till end of study, up to 12 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stiolto® Respimat® | ICS Plus LABA Plus LAMA (Triple Therapy)
Number analyzed (Participants) | 348 | 354
Months | NA [NA to NA] — Non-calculable as the median was not reached (and neither was the Q1). | NA [NA to NA] — Non-calculable as the median was not reached (and neither was the Q1).
Statistical Analysis 1: Comparison: Stiolto® Respimat® vs ICS Plus LABA Plus LAMA (Triple Therapy); Test type: Other; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.62 to 2.00] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Annual Rate of Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: Annual rate of severe chronic obstructive pulmonary disease (COPD) exacerbations.
  Severe exacerbation was a patient requiring hospitalization or emergency room visit due to COPD (ICD-9-491.21 or ICD-10-J44.1).
  Annual rate analysis utilized a negative binomial model with fixed effect of treatment (Stiolto Respimat versus triple therapy), logarithm of observational time as offset, and baseline prior ICS was used as a covariate.
Time Frame: Baseline till end of study, up to 12 months.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Arm/Group | Stiolto® Respimat® | Triple Therapy
Number analyzed (Participants) | 348 | 354
Exacerbations per participant per year | 0.07 [0.04 to 0.12] | 0.07 [0.04 to 0.11]
Statistical Analysis 1: Comparison: Stiolto® Respimat® vs Triple Therapy; Test type: Other; adjusted annual rate ratio = 1.08, 95% CI 2-sided [0.58 to 2.01] — Ratio: Stiolto Respimat/triple therapy

5. Secondary Outcome: Number of Patients With Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Over the 12 Month Observation Period
Description: Number of patients with moderate or severe chronic obstructive pulmonary disease (COPD) exacerbations over the 12 month observation period.
  Moderate exacerbation was a patient receiving an exacerbation-related prescription such as oral corticosteroid (prednisone or prednisolone) and/or antibiotic, but not requiring hospitalization.
  Severe exacerbation was a patient requiring hospitalization or emergency room visit due to COPD (ICD-9-491.21 or ICD-10-J44.1).
Time Frame: 12 months after baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stiolto® Respimat® | Triple Therapy
Number analyzed (Participants) | 348 | 354
Participants | 73 | 62
Statistical Analysis 1: Comparison: Stiolto® Respimat® vs Triple Therapy; A Cochran-Mantel-Haenszel (CMH) model with baseline ICS prior use as stratum was used to estimate the Risk Ratio (RR) (Stiolto Respimat versus triple therapy) of moderate or severe COPD exacerbations along with 95% CI; Test type: Other; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.89 to 1.64] — Ratio: Stiolto Respimat/triple therapy
Statistical Analysis 2: Comparison: Stiolto® Respimat® vs Triple Therapy; A Cochran-Mantel-Haenszel (CMH) model with baseline ICS prior use as stratum was used to estimate the Risk Difference (Stiolto Respimat versus triple therapy) of moderate or severe COPD exacerbations along with 95% CI; Test type: Other; Risk Difference (RD) = 0.036, 95% CI 2-sided [-0.022 to 0.094] — Ratio: Stiolto Respimat/triple therapy

ADVERSE EVENTS:
Time Frame: Up to 12 months + 21 days.
Description: All-Cause Mortality: all randomized patients allocated to original randomized treatment group. 5 patients in each group received the wrong prescription, these were included in the actual treatment.
  Adverse events (AE): all randomized patients who received a prescription of any study treatment.
  Non-serious AE collection and reporting was limited to events leading to trial discontinuation, treatment discontinuation or death as this is an approved product with a known safety profile.
Arm/Group | Stiolto® Respimat® | ICS Plus LABA Plus LAMA (Triple Therapy)
All-Cause Mortality (participants affected / at risk) | 12/356 | 12/358
Serious Adverse Events (participants affected / at risk) | 56/325 | 45/318
Other Adverse Events (participants affected / at risk) | 0/325 | 0/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stiolto® Respimat® (N=325) | ICS Plus LABA Plus LAMA (Triple Therapy) (N=318)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 1
Cardiac failure (Cardiac disorders) | 1 | 3
Cardiac failure acute (Cardiac disorders) | 3 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0
Left ventricular failure (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 2 | 2
Generalised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 4 | 1
Influenza (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 9
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 3
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract infection viral (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Blood osmolarity decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 5 | 2
Heart rate increased (Investigations) | 2 | 0
Troponin increased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 20 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Transcatheter aortic valve implantation (Surgical and medical procedures) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03265145/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03265145/SAP_001.pdf